CLINICAL TRIAL: NCT01247194
Title: A Phase 1b Study to Assess the Safety, Antiviral Efficacy and Pharmacokinetics of PPI-461 in Patients With HCV Genotype-1 Infection
Brief Title: A Phase 1b Study of PPI-461 in Patients With HCV Genotype 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Presidio Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPI-461-102; 2010-021510-36 (EudraCT Number)
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Genotype 1 Hepatitis C Virus Infection
Keywords: hepatitis C; NS5A; HCV RNA
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A (Active Comparator): PPI-461 50 mg
  or placebo
  Interventions: Drug: PPI-461; Drug: Placebo
- Cohort B (Active Comparator): PPI-461 100 mg
  or placebo
  Interventions: Drug: PPI-461; Drug: Placebo
- Cohort C (Active Comparator): PPI-461 200 mg
  or placebo
  Interventions: Drug: PPI-461; Drug: Placebo

INTERVENTIONS:
Drug: PPI-461 — capsule, oral, once daily for 3 days
Drug: Placebo — capsules, oral, once daily for 3 days

SUMMARY:
The purpose of the study is to assess the safety, tolerability, antiviral effects, and pharmacokinetics of PPI-461 in patients with chronic hepatitis C virus genotype 1 infection.

ELIGIBILITY:
Eligibility Criteria:

* Male or female, between 18 and 65 years of age (female patients must be surgically sterile or 2 years post-menopausal and are required to take a pregnancy test)
* Body Mass Index (BMI) 18 - 32 kg/m2
* Chronically infected with hepatitis C genotype-1 virus
* Serum HCV RNA > 5 log10 IU/mL
* No previous treatment with interferon, peginterferon, ribavirin or any investigational HCV antiviral agents
* No history of signs or symptoms of decompensated liver disease
* No known history of cirrhosis
* No co-infection with HBV, HIV-1, HIV-2
* No history of any medical condition that may interfere with absorption, distribution or elimination of study drug or with the clinical and laboratory assessments in this study
* No history of alcohol abuse, or illicit drug use within 2 years prior to Screen, or enrollment in a methadone maintenance program (unless he/she has been enrolled in the methadone program for at least 3 months with good compliance, stable psychosocial circumstances, and no known current risks for recidivism)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, as measured by clinical adverse events and laboratory assessments | up to Study Day 16 (14 days after the last PPI-461 dose)
Antiviral effects of PPI-461, as measured by HCV RNA levels | Up to Study Day 16 (14 days after the last PPI-461 dose)
PPI-461 pharmacokinetics as measured by plasma PPI-461 concentrations | Up to Study Day 10 (8 days after the last PPI-461 dose)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Brown, M.D., Study Director — Presidio Pharmaceuticals
Locations (9):
- United States (2):
  - Local Institution, Sacramento, California
  - Local institution, San Francisco, California
- Denmark (6):
  - Local institution, Aarhus
  - Local institution, Copenhagen
  - Local institution, Herlev
  - Local institution, Hvidovre
  - Local institution, Kolding
  - Local institution, Odense
- Local institution, London, United Kingdom